CLINICAL TRIAL: NCT03360682
Title: Pilot Single-Arm Clinical Trial to Evaluate the Efficacy, PK Interactions and Safety of Dolutegravir Plus 2 NRTIs in HIV-1-Infected Solid Organ Transplant Patients
Brief Title: Clinical Trial to Evaluate the Efficacy, Pharmacokinetics (PK) Interactions and Safety of Dolutegravir Plus 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs) in HIV-1-Infected Solid Organ Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTG-SOT; 2017-000469-62 (EudraCT Number)
Record Dates: First submitted 2017-10-30; First posted 2017-12-04 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HIV-1-infection; Solid Organ Transplant
MeSH Terms: interventions — Lamivudine; abacavir; dolutegravir; Tenofovir; Tablets; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-1-infected solid organ transplant patients 1 (Experimental): The patient or donor is not a carrier of genetic characteristics that predispose to a severe allergy to Abacavir or the patient is not a carrier of the hepatitis B virus.
  treatment 48 weeks
  Interventions: Drug: Lamivudine 300 MG; Drug: Abacavir 600 MG; Drug: Dolutegravir 50 mg
- HIV-1-infected solid organ transplant patients 2 (Experimental): The patient or donor is a carrier of genetic characteristics that predispose to a severe allergy to Abacavir or the patient is a carrier of the hepatitis B virus.
  treatment 48 weeks
  Interventions: Drug: Dolutegravir 50 mg; Drug: Tenofovir Disoproxil 245Mg Tablet; Drug: Emtricitabine 200 MG

INTERVENTIONS:
Drug: Lamivudine 300 MG — Lamivudine 300 MG/day (48 weeks)
  Other Names: J05AF05
  Arms: HIV-1-infected solid organ transplant patients 1
Drug: Abacavir 600 MG — Abacavir 600 MG/day (48 weeks)
  Other Names: J05AF06
  Arms: HIV-1-infected solid organ transplant patients 1
Drug: Dolutegravir 50 mg — Dolutegravir 50 MG/day (48 weeks)
  Other Names: J05AX12
Drug: Tenofovir Disoproxil 245Mg Tablet — Tenofovir 245 MG/day (48 weeks)
  Other Names: J05AF07
  Arms: HIV-1-infected solid organ transplant patients 2
Drug: Emtricitabine 200 MG — Emtricitabine 200 MG/day (48 weeks)
  Other Names: J05AF09
  Arms: HIV-1-infected solid organ transplant patients 2

SUMMARY:
The aims of this study are to obtain pharmacokinetic data on interactions between dolutegravir (DTG) and immunosuppressant drugs (Cyclosporine A, Tacrolimus, Sirolimus and Mycophenolic acid) in solid organ transplant (SOT) recipients to provide proof of principle data that DTG plus 2 nucleosides (NUCs) is safe and effective in HIV-infected SOT recipients.

ELIGIBILITY:
Inclusion Criteria:

1. HIV patients >18 years old who provide signed and dated informed consent;
2. Males and females;
3. SOT recipients (heart, liver or kidney);
4. On stable antiretroviral therapy (ART) for ≥6 months preceding the screening visit;
5. Plasma HIV RNA <50 cop/ml for 12 months (2 tests separated by at least 12 months with no viral load >50 between determinations);
6. Absence of major reverse transcriptase or integrase gene mutations affecting study drug efficacy by proviral DNA sequencing

Exclusion Criteria:

1. HIV patients who have stopped ART due to virological failure;
2. HIV patients who require treatment with DTG contraindicated medications;
3. History or presence of an allergy or intolerance to the study drug;
4. Active opportunistic infection;
5. Neoplasms requiring chemotherapy.
6. Pregnancy or breast feeding or planned pregnancy during the study period
7. Any other contraindication to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Miró Meda, MD, Principal Investigator — Hospital Clínico y provincial de Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PMCID: PMC12007624 — https://pubmed.ncbi.nlm.nih.gov/40256046/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: HIV-1-infected adults (>18) with kidney, liver, or heart transplant, on stable ART ≥6 months, HIV RNA <50 c/mL for 12 months, no major resistance mutations, and HLA-B*5701 negative.
  Some participants had switched to DTG + 2 NRTIs within the 48 weeks prior to study inclusion, while others switched at the time of enrollment. All participants were followed for 48 weeks from the start of DTG-based ART.
Groups:
- DTG + 2 NRTIs: Dolutegravir plus 2 NRTIs in HIV-1-infected solid organ transplant recipients
Period: Overall Study
Arm/Group | DTG + 2 NRTIs
Started | 19
Completed | 16
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | DTG + 2 NRTIs
Number analyzed (Participants) | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [51 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race and ethnicity data were not collected as part of this study.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Pharmacokinetic Parameters (Cmax, Cmin) of CsA Immunosuppressant
Description: Change in pharmacokinetic parameters (Cmax, Cmin) of immunosuppressant Cyclosporine A (CsA)
Time Frame: 24-hours before the switch and 24-hours 2 weeks after switching
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Pharmacokinetic (PK) Subset Before ART Change; Pharmacokinetic (PK) Subset After 2wk ART Change: Sub-group analysis
Arm/Group | Pharmacokinetic (PK) Subset Before ART Change | Pharmacokinetic (PK) Subset After 2wk ART Change
Number analyzed (Participants) | 2 | 2
ng/mL
  Cmax | 825 [686 to 946] | 299 [120 to 478]
  Cmin | 86.5 [83 to 90] | 98.5 [65 to 132]

2. Secondary Outcome: Viral Resistance
Description: number op patients with VIH viral load > 50 copies/mL virological failure.
Time Frame: week 48
Reporting Status: Not Posted

3. Secondary Outcome: Changes in CD4+ Cell
Description: To assess the changes in CD4+ cell count >200 cel/mL in peripheral blood.
Time Frame: week 48
Reporting Status: Not Posted

4. Secondary Outcome: Lipid Profile
Description: To assess the changes in lipid profile (triglycerides)
Time Frame: week 48
Reporting Status: Not Posted

5. Secondary Outcome: Renal Function
Description: To assess creatinine >normal valors mg/dl> 120 mg/dl
Time Frame: week 48
Reporting Status: Not Posted

6. Secondary Outcome: Safety: Number AEs and SAEs
Description: number AEs and SAEs
Time Frame: week 48
Reporting Status: Not Posted

7. Primary Outcome: Change in Pharmacokinetic Parameters (Cmax, Cmin) of MPA Immunosuppressant
Description: Change in pharmacokinetic parameters (Cmax, Cmin) of immunosuppressant Mycophenolic Acid (MPA).
Time Frame: 24-hours before the switch and 24-hours 2 weeks after switching
Measure: Median (Inter-Quartile Range); unit: μg/mL
Arm/Group | Pharmacokinetic (PK) Subset Before ART Change | Pharmacokinetic (PK) Subset After 2wk ART Change
Number analyzed (Participants) | 7 | 7
μg/mL
  Cmax | 6.3 [3.8 to 10.7] | 10.3 [5.3 to 12.9]
  Cmin | 1.9 [1.5 to 2.5] | 2.9 [1.7 to 4]

8. Primary Outcome: Change in Pharmacokinetic Parameters (Cmax, Cmin) of Tacrolimus Immunosuppressant
Time Frame: 24-hours before the switch and 24-hours 2 weeks after switching
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pharmacokinetic (PK) Subset Before ART Change | Pharmacokinetic (PK) Subset After 2wk ART Change
Number analyzed (Participants) | 7 | 7
ng/mL
  Cmax | 14.4 [10.8 to 18.3] | 16.4 [12.1 to 18.7]
  Cmin | 6.2 [5.2 to 8.9] | 4.4 [4.3 to 8.5]

ADVERSE EVENTS:
Time Frame: Up to 48 weeks of treatment plus 28 days after last dose in case of early withdrawal.
Description: Only adverse events leading to treatment discontinuation or considered clinically relevant are reported individually. All other AEs occurred with low frequency and were not considered related to treatment.
Arm/Group | DTG + 2 NRTIs
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 2 NRTIs (N=19)
Cytomegalovirus infection (Infections and infestations) | 1 (1) — Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 2 NRTIs (N=19)
Insomnia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety symptoms (Nervous system disorders) | 1 (1)
Other (General disorders) | 10 (10)
Hyperglycemia (Endocrine disorders) | 1 (1) — With difficult medical control
Diarrhea (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was a single-arm pilot trial with a small sample size, which may limit generalizability. The number of participants included in the pharmacokinetic analysis of cyclosporine A was limited, and therefore insufficient to support robust statistical conclusions. No control group was included, and all participants received DTG-based ART. Further studies are needed to confirm findings in larger cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03360682/Prot_SAP_000.pdf